CLINICAL TRIAL: NCT06178445
Title: Efficacy and Safety of GemCis Plus Trastuzumab Plus Pembrolizumab in Previously Untreated HER2-positive Biliary Tract Cancer
Acronym: TRAP-BTC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Medizinische Hochschule Hannover, Germany, Prof. Dr. Arndt Vogel (Unknown); MSD Sharp & Dohme GmbH, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAP-BTC; EU CT number (Other: European Union)
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer; HER2 Gene Mutation; HER2
Keywords: cholangiocarcinoma; gallbladder carcinoma; HER2-positive; HER2
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Trastuzumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: All eligible patients will receive SOC treatment with gemcitabine/cisplatin in combination with trastuzumab and pembrolizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SOC treatment with gemcitabine/cisplatin in combination with trastuzumab and pembrolizumab (Experimental): * Gemcitabine: 1000 mg/m2 on day 1 and day 8 of each 21-days cycle (Q3W)
  * Cisplatin: 25 mg/m2 on day 1 and day 8 of each 21-days cycle
  * Trastuzumab: initial dose 8 mg/kg, then 6 mg/kg on day 1 of each 21-days cycle
  * Pembrolizumab: 200 mg on day 1 of each 21-days cycle
  Interventions: Drug: SOC plus trastuzumab and pembrolizumab

INTERVENTIONS:
Drug: SOC plus trastuzumab and pembrolizumab — SOC treatment with gemcitabine/cisplatin in combination with trastuzumab and pembrolizumab

SUMMARY:
This is a multicenter, single arm, prospective, open-label phase II trial investigating the clinical activity triplet regimen consisting of a combination of chemotherapy (gemcitabine/cisplatin) + trastuzumab + pembrolizumab as first-line treatment for cholangiocarcinoma and gallbladder cancer patients.

Patients suffering from previously untreated HER2 (human epidermal growth factor receptor 2) positive, unresectable cholangiocarcinoma and gallbladder cancer will be included in the study and are scheduled to receive triplet regimen consisting of a combination of pembrolizumab, trastuzumab and gemcitabine/cisplatin (GemCis).

ELIGIBILITY:
Inclusion Criteria:

1. Participant provides written informed consent.
2. Male/female Participants who are at least 18 years of age on the day of signing informed consent.
3. Participant is, in the investigator's judgement, willing and able to comply with the study protocol.
4. Participant has histologically confirmed diagnosis of cholangiocarcinoma or gallbladder cancer.
5. Participant is not eligible for surgery.
6. Participants must have HER2-positive disease defined as either IHC 3+ or IHC 2+, the latter in combination with FISH+, as assessed locally on primary tumor OR positively confirmed by NGS-analysis OR positively confirmed by mRNA
7. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
8. Male Participants must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 7 months after the last dose of study treatment and refrain from donating sperm during this period.

   Female Participants are eligible to participate if they are not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   * Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   * A WOCBP who agrees to follow the contraceptive guidance as given in Appendix 3 during the treatment period and for at least 7 months after the last dose of study intervention
9. Participant has measurable disease based on RECIST v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
10. Have adequate organ function as defined in the following table (Table 2).
11. Criteria for known Hepatitis B and C positive subjects Hepatitis B and C screening tests are not required unless there is a known history of HBV or HCV infection and/or as mandated by local health authority

    1. Hepatitis B positive subjects

       * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load (< 100 IU/mL) prior to enrollment
       * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
    2. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

       * Participants must have completed curative anti-viral therapy at least 4 weeks prior to enrollment.

Exclusion Criteria:

1. Participant has received prior systemic anti-cancer therapy NOTE: Participants who have received up to 4 cycles of prior GemCis or any other anti-cancer treatment prior to initiation of study treatment are eligible for the study. In case of other anti-cancer treatment, at study inclusion patients must be switched to study treatment as defined in protocol section 5.2.
2. Participant has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).

   NOTE: Up to 4 cycles of prior anti-cancer therapy are allowed. In case of other anti-cancer treatment, at study inclusion patients must be switched to study treatment as defined in protocol section 5.2.
3. Participant has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Participant has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
5. Participant is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   NOTE: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Participant has known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
8. Participant has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
9. Participant has severe hypersensitivity (≥grade 3) to pembrolizumab, trastuzumab, gemcitabine, cisplatin and/or any of their excipients.
10. Participant has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
11. Patient has inadequate cardiac function (LVEF value < 55%) as determined by echocardiography.
12. Participant has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Participant has an active infection requiring systemic therapy.
14. Participant has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Participant has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Participant has had an allogenic tissue/solid organ transplant.
17. Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Participants who are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 7 months after the last dose of trial treatment.
19. Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan, previous allogenic bone marrow/blood transplantation or any psychiatric disorder or substance abuse that prohibits obtaining informed consent
20. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
21. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].
22. Patients who are dependent on the sponsor, the investigator or the trial site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  defined as proportion of subjects with complete response (CR) or partial response (RP) according to unconfirmed RECIST v1.1 at 6 months after treatment initiation

SECONDARY OUTCOMES:
PFS | through study completion, an average of 2 years
  defined as time from enrolment until the date of first objectively documented progression according to RECIST v1.1
OS | through study completion, an average of 2 years
  defined as time from enrolment to the date of death of any cause
PFS rate at 6 months | 6 months
  defined as proportion of patients without progression after 6, 9 and 12 months
PFS rate at 9 months | 9 months
  defined as proportion of patients without progression after 9 months
PFS rate at 12 months | 12 months
  defined as proportion of patients without progression after 12 months
The incidence, nature, causality, seriousness, and severity of adverse events using NCI CTCAE 5.0 | through study completion, an average of 2 years
  Safety of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Frankfurter Institut fuer Klinische Krebsforschung IKF GmbH
Locations (7):
- Germany (7):
  - Charité Universitätsmedizin, Berlin
  - Krankenhaus Nordwest (KHNW), Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Göttingen, Göttingen
  - Hämatologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - LMU München, München

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared